CLINICAL TRIAL: NCT03845920
Title: Modulation of Cognitive Flexibility by Transcranial Direct Current Stimulation, Tyrosine Administration and Polymorphisms in the COMT Gene
Brief Title: Mod of Cognitive Flexibility by tDCS, Tyrosine Polymorphisms in the COMT Gene
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SheffieldHallamAquili2019
Record Dates: First submitted 2019-02-11; First posted 2019-02-19 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Modulation of Cognitive Flexibility by Transcranial Direct Current Stimulation, Tyrosine Administration and Polymorphisms in the COMT Gene
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Pharmaceutical Preparations; Tyrosine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tDCS sham + placebo (Other): tDCS= transcranial direct current stimulation drugs= placebo (cellulose [2 grams])
  Interventions: Combination Product: tdcs (sham/anodal) + drug (placebo/tyrosine)
- tDCS sham + tyrosine (Experimental): tDCS= transcranial direct current stimulation drugs= tyrosine (2 grams)
  Interventions: Combination Product: tdcs (sham/anodal) + drug (placebo/tyrosine)
- tDCS anodal + placebo (Experimental): tDCS= anodal transcranial direct current stimulation of the dorsolateral prefrontal cortex drugs= placebo (cellulose [2 grams])
  Interventions: Combination Product: tdcs (sham/anodal) + drug (placebo/tyrosine)
- tDCS anodal +tyrosine (Experimental): tDCS= anodal transcranial direct current stimulation of the dorsolateral prefrontal cortex drugs= tyrosine (2 grams)
  Interventions: Combination Product: tdcs (sham/anodal) + drug (placebo/tyrosine)

INTERVENTIONS:
Combination Product: tdcs (sham/anodal) + drug (placebo/tyrosine) — tDCS= A DC Stimulator Plus (neuroConn, Germany) with one 5 cm x 7 cm rubber electrode (anode) and a 10 cm x 10 cm (cathode; reference electrode), encased in saline soaked sponges will be used. The anode will be positioned over the left dlPFC, centered on F3 in the 10e20 electroencephalography (EEG) system, while the cathode on the contralateral supraorbital ridge (Fp2).Current will be delivered at 1.5mA for 20 min plus 30 s fade in/fade out periods.For sham stimulation, the current will be faded in over 30 s, at 1.5mA and then will be switched off.
  Drugs= 2.0 g of L-Tyrosine and 2.0 g of the placebo microcrystalline cellulose will be dissolved in 400ml of orange juice as per previously published protocols.

SUMMARY:
The current study would examine whether increases in endogenous dopaminergic activity via tyrosine and the (presumed) excitation of these by anodal tDCS of the dlPFC could causally be related to cognitive flexibility as measured by task switching and reversal learning.

Additionally, the study will test whether the Val158Met-polymorphism in the catechol- O-methyltransferase (COMT) gene could also predict the effect of TYR supplementation, as this gene is involved in DA degradation in the prefrontal cortex.

ELIGIBILITY:
Inclusion Criteria:

* • Either male or female

  * Between 18 and 30 years
  * You are in good health
  * You agree to fast overnight prior to testing

Exclusion Criteria:

* • Are suffering from cardiac, hepatic, renal, neurological disorders

  * Damaged or diseased skin on your face and scalp, or a sensitive scalp
  * A history of alcohol or drug addiction, or severe psychiatric illness
  * Drug treatment which may lower seizure threshold (i.e. epilepsy)
  * Pregnancy
  * Sleep deprivation (less than 6 hours a day)
  * A history of migraine or headaches
  * A history of taking antidepressants
  * A history of taking tyrosine supplements

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Wisconsin Card Sorting Test (WCST) performance | Measured twice in each session (4 arms): at time 0 and 80 minutes into testing.
  Measuring change in perseverative errors in the WCST
Probabilistic Reversal Learning (PRL) performance | Measured twice in each session (4 arms): at time 0 and 80 minutes into testing.
  Measuring change in reversal errors in the WCST
Flanker Task performance | Measured twice in each session (4 arms): at time 0 and 80 minutes into testing.
  Measuring change in conflict cost (defined as the difference in reaction time between congruent and incongruent responses)

CONTACTS AND LOCATIONS:
Overall Officials: Luca Aquili, Ph.D., Principal Investigator — Sheffield Hallam University
Locations (1):
- Psychology labs, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No